CLINICAL TRIAL: NCT01692574
Title: Treatment of Obesity in Depressed Individuals: A Randomized Controlled Trial
Brief Title: Treatment for Depressed, Obese Individuals at Risk for Cardiovascular Disease (CVD)
Acronym: TODI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 813829
Record Dates: First submitted 2012-09-20; First posted 2012-09-25 (Estimated); Last update posted 2016-08-22 (Estimated); Status verified 2016-08

CONDITIONS: Obesity; Major Depressive Disorder; Dysthymic Disorder; Cardiovascular Disease
Keywords: depression and obesity treatment
MeSH Terms: conditions — Obesity; Depressive Disorder, Major; Dysthymic Disorder; Cardiovascular Diseases; Depression | interventions — Behavior Therapy; Cognitive Behavioral Therapy; Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Combined (Experimental): Group cognitive-behavior therapy for depression combined with behavior modification for weight loss
  Interventions: Behavioral: Behavior Modification for Weight Loss; Behavioral: Cognitive-Behavior Therapy for Depression
- GCBT-ND (Active Comparator): Group cognitive-behavior therapy for depression combined with an alternative approach to weight loss
  Interventions: Behavioral: Alternative Approach to Weight Loss; Behavioral: Cognitive-Behavior Therapy for Depression
- DSE (Active Comparator): Behavior modification for weight loss combined with depression support and education.
  Interventions: Behavioral: Behavior Modification for Weight Loss; Behavioral: Depression Support and Education

INTERVENTIONS:
Behavioral: Behavior Modification for Weight Loss
  Arms: Combined; DSE
Behavioral: Alternative Approach to Weight Loss
  Arms: GCBT-ND
Behavioral: Cognitive-Behavior Therapy for Depression
  Arms: Combined; GCBT-ND
Behavioral: Depression Support and Education
  Arms: DSE

SUMMARY:
To determine whether individuals who suffer from depression and obesity are able to lose weight and show improvements in mood and cardiovascular disease risk factors following 20 weeks of a combined treatment of cognitive-behavior therapy for depression and behavior modification for weight loss. Participants will be assigned to one of three treatments: 1) cognitive-behavior therapy for the treatment of depression combined with an alternative approach to weight loss, 2) a weight loss intervention combined with a depression support and education , or 3) cognitive-behavioral therapy for depression combined with a weight loss intervention.

ELIGIBILITY:
Inclusion Criteria

* Female and male participants, with a BMI of 27 kg/m2 to 45 kg/m2
* Age 18 - 70 years old
* Presence of current major depressive disorder or dysthymic disorder
* At least 2 CVD risk factors, as characterized by the metabolic syndrome, including:

  * Elevated waist circumference (males 40 inches or 102 cm; females 35 inches of 88 cm)
  * Fasting blood glucose 100 mg/dL
  * Blood pressure 130/85 mm Hg
  * Triglycerides 150 mg/dL
  * Reduced HDL cholesterol (males 40 mg/dL; females 50 mg/dL)
  * OR medications for these conditions
* Able to comply will all study procedures and schedule
* Able to speak and read English

Exclusion Criteria

* Cardiovascular event (e.g., myocardial infarction, stroke) within the past 12 months
* Use of tricyclic anti-depressants, monoamine oxidase inhibitors or paroxetine, mood stabilizers, or antipsychotic medications. (Note: participants who take SSRI/SNRI may be acceptable, provided they have been on a stable dose of these medications 3 months.)
* Use of weight-loss medications or any medications known to significantly affect weight (e.g., oral steroids) in past 3 months
* Weight loss of 5% or more in past 6 months
* Enrollment in weight reduction program in prior 3 months
* Treatment in individual psychotherapy for any psychiatric disorder in prior 3 months (Note: participants in couples or family counseling will be allowed.)
* Severe depression or severe impairment of functioning as judged by the assessor or PI
* Presence of active suicidal ideation
* Diabetes
* Alcohol/drug abuse/dependence
* Renal/hepatic disease
* Change in thyroid medications in last 3 months
* Pregnant/lactating, within 6-months post-partum
* Current diagnoses, or history within the last 5 years, of anorexia or bulimia
* Psychotic symptoms or hospitalization for a psychiatric disorder in previous 12 months
* Mood disorder NOS, substance-induced mood disorders, mood disorders due to a general medical condition
* History of bipolar disorder
* History of head trauma
* Any changes in smoking behavior in prior 3 months (or plans to change in the next 3 months)
* Plans for bariatric surgery
* Any other uncontrolled major medical problems
* Women who are pregnant

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2012-08; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Weight loss | Baseline to 20 weeks of treatment, follow-up at week 46
  To determine whether depressed, obese individuals who receive the combined treatment of cognitive-behavior therapy for depression and behavior modification for weight loss are able to lose 5% of their initial weight at the end of 20 weeks of treatment.

SECONDARY OUTCOMES:
Changes in metabolic cardiovascular disease risk factors and inflammatory markers | Baseline to 20 weeks of treatment, follow up at week 46

OTHER OUTCOMES:
Changes in mood | Baseline to 20 weeks of treatment, follow up at week 46

CONTACTS AND LOCATIONS:
Overall Officials: Lucy F Hemsley-Faulconbridge, PhD, Principal Investigator — University of Pennsylvania Center for Weight and Eating Disorders
Locations (1):
- University of Pennsylvania: Center for Weight and Eating Disorders, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Faulconbridge LF, Driscoll CFB, Hopkins CM, Bailer Benforado B, Bishop-Gilyard C, Carvajal R, Berkowitz RI, DeRubeis R, Wadden TA. Combined Treatment for Obesity and Depression: A Pilot Study. Obesity (Silver Spring). 2018 Jul;26(7):1144-1152. doi: 10.1002/oby.22209. PMID 29932516